CLINICAL TRIAL: NCT02742779
Title: A Phase I, Randomized, Single and Multiple Ascending Dose, Placebo-Controlled, Double-Blind Study to Determine the Safety, Tolerability, and Pharmacokinetics of GDC-0310 in Healthy Volunteers
Brief Title: A Study to Determine the Safety, Tolerability, and Pharmacokinetics of GDC-0310 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GN29829
Record Dates: First submitted 2016-03-11; First posted 2016-04-19 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (10):
- High-Fat Meal SD Cohort: PIC (Part 1) (Experimental): Participants will receive GDC-0310 single ascending dose based on PK results from earlier SD cohorts up to an established dose yielding at least a 2-fold exposure margin to the MTD administered orally following a high-fat meal after a 8-hour/overnight fast using PIC on Day 1 of the treatment period (5 days) in an additional cohort of Part 1.
  Interventions: Drug: GDC-0310
- High-Fat Meal SD Cohort: Solution Formulation (Part 3) (Experimental): Participants will receive GDC-0310 single ascending dose based on PK results from earlier SD cohorts up to an established dose yielding at least a 2-fold exposure margin to the MTD administered orally following a high-fat meal after a 8-hour/overnight fast using solution on Day 1 of the treatment period (5 days) in an additional cohort of Part 3.
  Interventions: Drug: GDC-0310
- Low-Fat Meal SD Cohort: PIC (Part 1) (Experimental): Participants will receive GDC-0310 single ascending dose given orally using PIC based on PK results from earlier SD cohorts up to an established dose yielding at least a 2-fold exposure margin to the MTD administered orally following a low-fat meal after an 8-hour/overnight fast using PIC on Day 1 of the treatment period (5 days) in an additional cohort of Part 1.
  Interventions: Drug: GDC-0310
- Low-Fat Meal SD Cohort: Solution Formulation (Part 3) (Experimental): Participants will receive GDC-0310 single ascending dose given orally using PIC based on PK results from earlier SD cohorts up to an established dose yielding at least a 2-fold exposure margin to the MTD administered orally following a low-fat meal after an 8-hour/overnight fast using solution on Day 1 of the treatment period (5 days) in an additional cohort of Part 1.
  Interventions: Drug: GDC-0310
- MD Cohort: PIC (Part 2) (Experimental): Participants will receive multiple ascending dose administered orally using PIC from Day 1 to Day 13 twice daily (BID) or may even be thrice daily (TID) or four times a day (QD) depending on clinical PK, followed by morning dose on Day 14 in 7 cohorts of Part 2.
  Interventions: Drug: GDC-0310
- MD Cohort: Solution Formulation (Part 4) (Experimental): Participants will receive multiple ascending dose in fed or fast condition, administered orally using solution from Day 1 to Day 13 BID or may even be TID or QD depending on clinical PK, followed by morning dose on Day 14 in 7 cohorts of Part 2.
  Interventions: Drug: GDC-0310
- Placebo PIC (Placebo Comparator): Participants will receive placebo matched to GDC-0310 single or multiple ascending dose administered orally in the fasted (SD cohorts) or fed state using PIC on Day 1 of the treatment period (5 days) to the SD cohorts and from Day 1 to 14 BID or may even be TID or QD depending on clinical PK, to the MD cohorts.
  Interventions: Drug: Placebo
- Placebo Solution (Placebo Comparator): Participants will receive placebo matched to GDC-0310 single or multiple ascending dose administered orally in the fasted (SD cohorts) or fed state using PIC on Day 1 of the treatment period (5 days) to the SD cohorts and from Day 1 to 14 BID or may even be TID or QD depending on clinical PK, to the MD cohorts.
  Interventions: Drug: Placebo
- SD Cohort: PIC (Part 1) (Experimental): Participants will receive GDC-0310 single ascending dose administered orally in the fasted state using PIC on Day 1 of the treatment period (5 days) in the 9 cohorts of Part 1.
  Interventions: Drug: GDC-0310
- SD Cohort: Solution Formulation (Part 3) (Experimental): Participants will receive GDC-0310 single ascending dose administered orally in the fasted state using solution formulation on Day 1 of the treatment period (5 days) in the 9 cohorts of Part 3.
  Interventions: Drug: GDC-0310

INTERVENTIONS:
Drug: GDC-0310 — Participants will receive single or multiple ascending doses of GDC-0310 orally in fasted or fed state.
  Arms: High-Fat Meal SD Cohort: PIC (Part 1); High-Fat Meal SD Cohort: Solution Formulation (Part 3); Low-Fat Meal SD Cohort: PIC (Part 1); Low-Fat Meal SD Cohort: Solution Formulation (Part 3); MD Cohort: PIC (Part 2); MD Cohort: Solution Formulation (Part 4); SD Cohort: PIC (Part 1); SD Cohort: Solution Formulation (Part 3)
Drug: Placebo — Participants will receive placebo matched to GDC-0310 as single or multiple oral dose in fasted or fed state.
  Arms: Placebo PIC; Placebo Solution

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple orally ascending doses of GDC-0310 administered in healthy participants as 4 parts including Part 1- a single dose (SD) part using a powder-in-capsule (PIC) formulation, Part 2- a multiple dose (MD) part using a PIC formulation, Part 3- a SD part using a solution formulation, and Part 4- a MD part using a solution formulation. Effects of food on pharmacokinetics (PK) will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential must meet the criteria defined in the protocol
* Body mass index within the range of 18.0 to 30.0 kilograms per meter square (kg/m^2), inclusive, and a minimum weight of 50.0 kg

Exclusion Criteria:

* Have a clinically significant medical condition (e.g., hypertension; diabetes; impaired cardiac, renal or hepatic function; hyperthyroidism or hypothyroidism; neurological disorder; pain condition; hematologic disorder; psychiatric disorders requiring chronic medication) including any medical condition requiring treatment with medication (other than study drugs and medications specifically allowed by this protocol) during participation in the study
* Evidence of any hepatic impairment including any abnormal levels (i.e., greater than [>] 1 × the upper limit of normal) of alkaline phosphatase, gamma glutamyl transpeptidase, alanine transaminase, aspartate aminotransferase or bilirubin
* Evidence of clinically significant renal impairment defined as >1.3 × upper limit of normal creatinine
* History or presence of alcoholism or alcohol or substance abuse (not including nicotine or caffeine) within the previous 2 years or routinely consume 2 or more alcohol-containing beverages per day or more than 10 units of alcohol per week (1 unit =150 milliliter (mL) of wine, 360 mL of beer, or 45 mL of 40 percent (%) alcohol)
* Have a positive urine drug test at screening or check-in or any other point during the study
* Are habituated to analgesic drugs (i.e., routine use of oral analgesics 5 or more times per week) or have a history of chronic pain requiring opiate use
* Have used tobacco or nicotine-containing products within 3 months before study drug administration
* Have clinically significant abnormal laboratory values as determined by the principal investigator
* Have used any prescription or over-the-counter medication or supplement within 14 days or 5 times the elimination half-life (whichever is longer) before administration of study drug and until the end of their participation in the study
* History of seizures, including in first degree relatives
* History of heritable myopathy, weakness, or paralysis, including in first degree relatives indicative of familial periodic paralysis
* Current treatment with medications that are well known to prolong the QT interval

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs) | Baseline up to Month 9

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: Pre-dose (PD) (Hour[H] 0),5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H post-dose(PoD); MD Cohort:PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14;Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Minimum Plasma Concentration (Cmin) of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Time to Maximum Plasma Concentration (tmax) of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Area Under the Concentration-Time Curve (AUC) of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Apparent Clearance (CL/F) of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Apparent Terminal Volume of Distribution (Vz/F) of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Apparent Terminal Elimination Rate Constant (ke) of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Apparent Terminal Half-Life (t1/2) of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Pharmacokinetics (PK) Dose Proportionality as Assessed With Cmax of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
PK Dose Proportionality as Assessed With AUC of GDC-0310 | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  SD Cohort: PD H 0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16,24,48,96H PoD; MD Cohort: PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15
Accumulation Ratio for MD Cohort | Pre dose up to Day 15 (detailed timeframe has been reported in the description)
  PD H0,5 minutes,0.25,0.5,1,1.5,2,3,4,6,8,10,12,13,14,16H PoD on Day 1,14; Pre a.m. dose (H0) on Day 2,3,4,5,7,9,11,13;24H PoD on Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States